CLINICAL TRIAL: NCT03461107
Title: Evaluation of Beta-adrenergic Receptor Gene Polymorphisms in the Long-term Effects of Beta-blockade in Patients With Chronic Heart Failure
Brief Title: Evaluation of Clinical and Genetic Modifiers of Long-term Survival in Heart Failure
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Tongji Hospital (Other)
Responsible Party: Principal Investigator, Dao Wen Wang, Prof, Tongji Hospital
Other Study IDs: TJ-HF-ARB
Record Dates: First submitted 2018-03-05; First posted 2018-03-09 (Actual); Last update posted 2019-04-10 (Actual); Status verified 2019-04

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- patients with heart failure
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention

SUMMARY:
The purpose of this study is to evaluate the beta-adrenergic receptor gene polymorphisms in the long-term effects of beta-blockade in patients with chronic heart failure.

ELIGIBILITY:
Inclusion Criteria:

1. 18 years of age or older;
2. Patients are required to have chronic heart failure (NYHA II-IV) with a left ventricular ejection fraction lower than 40%;
3. Patients are voluntary and signed informed consent.

Exclusion Criteria:

1. Pregnant women or plan to;
2. Participate in any drug clinical trials within 3 months;
3. Serious neurological disease (Alzheimer's disease, Parkinson syndrome, progressive lower limbs or deaf patients);
4. Previous history of cancer or tumor, or pathological examination confirmed precancerous lesions;
5. Patients refused to comply with the requirements of this study to complete the research work;
6. According to the researchers, patients can not complete the study or not to comply with the requirements of this study (because of the reasons for the management or other reasons).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 2500 outpatients or hospitalized patients with chronic heart failure will be enrolled in this study.
Sampling Method: Non-Probability Sample
Enrollment: 2500 (Estimated)
Dates: Start 2016-04-18 (Actual); Primary Completion 2019-12-31 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
Cardiovascular death | up to 24 months
Heart transplantation | up to 24 months

SECONDARY OUTCOMES:
All cause death | up to 24 months
Heart failure recuring | up to 24 months
Readmission because of cardiovascular diseases | up to 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Dao Wen Wang, doctor, Principal Investigator — Tongji Hospital
Locations (1):
- Tongji Hospital, Wuhan, Hubei, China

REFERENCES:
- [Derived] Zhao C, Jiang X, Peng L, Zhang Y, Li H, Zhang Q, Wang Y, Yang F, Wu J, Wen Z, He Z, Shen J, Chen C, Wang DW. Glimepiride, a novel soluble epoxide hydrolase inhibitor, protects against heart failure via increasing epoxyeicosatrienoic acids. J Mol Cell Cardiol. 2023 Dec;185:13-25. doi: 10.1016/j.yjmcc.2023.10.009. Epub 2023 Oct 21. PMID 37871528
- [Derived] Zhao Y, Li H, Du H, Yin Z, He M, Fan J, Nie X, Sun Y, Hou H, Dai B, Zhang X, Cai Y, Jin K, Ding N, Wen Z, Chang J, Chen C, Wang DW. A Kaposi's sarcoma-associated herpes virus-encoded microRNA contributes to dilated cardiomyopathy. Signal Transduct Target Ther. 2023 Jun 9;8(1):226. doi: 10.1038/s41392-023-01434-3. PMID 37291118
- [Derived] Peng L, Song Z, Zhao C, Abuduwufuer K, Wang Y, Wen Z, Ni L, Li C, Yu Y, Zhu Y, Jiang H, Shen J, Jiang X, Chen C, Zhang X, Wang DW. Increased Soluble Epoxide Hydrolase Activity Positively Correlates with Mortality in Heart Failure Patients with Preserved Ejection Fraction: Evidence from Metabolomics. Phenomics. 2022 Oct 27;3(1):34-49. doi: 10.1007/s43657-022-00069-8. eCollection 2023 Feb. PMID 36939801
- [Derived] Wei H, Zhao M, Wu J, Li C, Huang M, Gao J, Zhang Q, Ji L, Wang Y, Zhao C, Dong E, Zheng L, Wang DW. Association of Systemic Trimethyllysine With Heart Failure With Preserved Ejection Fraction and Cardiovascular Events. J Clin Endocrinol Metab. 2022 Nov 25;107(12):e4360-e4370. doi: 10.1210/clinem/dgac519. PMID 36062477
- [Derived] Hu D, Xiao L, Li S, Hu S, Sun Y, Wang Y, Wang DW. Prediction of HF-Related Mortality Risk Using Genetic Risk Score Alone and in Combination With Traditional Risk Factors. Front Cardiovasc Med. 2021 Apr 26;8:634966. doi: 10.3389/fcvm.2021.634966. eCollection 2021. PMID 33981732
- [Derived] Hu D, Li S, Hu S, Sun Y, Xiao L, Li C, Wang J, Wang Y, Ni L, Zhao C, Wang DW. A Common Missense Variant in OMA1 Associated with the Prognosis of Heart Failure. Cardiovasc Drugs Ther. 2020 Jun;34(3):345-356. doi: 10.1007/s10557-020-06960-8. PMID 32236861
- [Derived] Hu D, Huang J, Hu S, Zhang Y, Li S, Sun Y, Li C, Cui G, Wang DW. A common variant of RIP3 promoter region is associated with poor prognosis in heart failure patients by influencing SOX17 binding. J Cell Mol Med. 2019 Aug;23(8):5317-5328. doi: 10.1111/jcmm.14408. Epub 2019 May 31. PMID 31148336